CLINICAL TRIAL: NCT04001829
Title: Prospective Validation Trial of Taxane Therapy (Docetaxel or Weekly Paclitaxel) and Risk of Chemotherapy-Induced Peripheral Neuropathy in African American Women
Brief Title: Taxane and Taxane-Induced Peripheral Neuropathy in African American Patients With Stage I-III Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EAZ171; NCI-2019-00266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAZ171 (Other: ECOG-ACRIN Cancer Research Group); ECOG-ACRIN-EAZ171 (Other: DCP); EAZ171 (Other: CTEP); UG1CA189828 (NIH)
Record Dates: First submitted 2019-06-19; First posted 2019-06-28 (Actual); Results first posted 2024-06-12 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Invasive Breast Carcinoma; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
Keywords: African American; Taxane; Docetaxel; Paclitaxel; TIPN; Neuropathy; Germline predictor; FCAMR GG genotype; SBF2 mutation
MeSH Terms: interventions — Docetaxel; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (paclitaxel) (Experimental): Patients receive paclitaxel IV over 3 hours once weekly. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients may also receive trastuzumab and/or pertuzumab per institution routine care per treating physician's discretion.
  Interventions: Drug: Paclitaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (docetaxel) (Experimental): Patients receive docetaxel IV over 1 hour once every 3 weeks. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity. Patients may also receive cyclophosphamide, doxorubicin, trastuzumab, and/or pertuzumab per institution routine care per treating physician's discretion.
  Interventions: Drug: Docetaxel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Arm B (docetaxel)
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm A (paclitaxel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies whether a prior germline predictor of taxane-induced peripheral neuropathy (TIPN) can help identify a subgroup of patients who are at higher risk of chemotherapy-induced peripheral neuropathy in African American patients with stages I-III breast cancer. The study also investigates whether docetaxel maybe work better than paclitaxel with regard to TIPN rate/severity and dose reductions.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Prospectively validate a prior germline predictor of TIPN using the Common Terminology Criteria for Adverse Events (CTCAE). Specifically, this study will demonstrate that patients with a high-risk TIPN genotype have significantly more grade 2-4 TIPN than patients with a low risk genotype.

SECONDARY OBJECTIVES:

I. Validate a prior germline predictor of TIPN using the Functional Assessment of Cancer Therapy (FACT)/Gynecologic Oncology Group (GOG)-Neurotoxicity (NTX) neurotoxicity subscale in Arm A.

II. Compare grade 2-4 TIPN based on CTCAE between weekly paclitaxel (Arm A) versus (vs.) every three-week docetaxel (Arm B).

III. Prospectively confirm dose reductions due to TIPN are lower for every three-week docetaxel compared with weekly paclitaxel in a prospective cohort of patients of African ancestry.

IV. Prospectively confirm dose reductions due to any cause are lower for every three-week docetaxel compared with weekly paclitaxel in a prospective cohort of patients of African ancestry.

V. Assess the ability of the high-risk genotype to predict TIPN risk for docetaxel.

EXPLORATORY OBJECTIVES:

Correlative Study Objectives:

I. Identify novel markers of TIPN and elucidate the mechanism. II. Whole genome sequencing of germline blood to evaluate for additional predictors of TIPN.

III. Create induced pluripotent stem cell (iPSC) derived neurons from patient samples.

IIIa. Evaluate whether clinical findings can be mimicked in vitro. IIIb. Evaluate gene expression (ribonucleic acid [RNA] sequencing [seq]) and the epigenome at baseline versus after exposure in those prone to TIPN versus those not.

IV. Create a biorepository of patient derived samples for future translational research.

Patient-Reported Outcome Objectives:

I. Compare Grade 2-4 TIPN (moderate to life threatening) based on Patient Reported Outcomes (PRO)-CTCAE items between weekly paclitaxel (Arm A) vs. every three-week docetaxel (Arm B).

II. Prospectively compare FACT/GOG-NTX Health-Related Quality of Life (HRQoL) subscale, Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function version (v.)2 Short Form (SF) 10a, scores between every three-week docetaxel and weekly paclitaxel and between high risk and low risk genotypes (Arm A) in a cohort of African ancestry.

III. Compare the impact on financial toxicity (Comprehensive Score for Financial Toxicity [COST] scores) for every three-week docetaxel compared with weekly paclitaxel.

IV. Examine associations between social determinants of health (zip code, marital status, education, income & insurance status) and dose reductions and treatment discontinuation.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM A: Patients receive paclitaxel intravenously (IV) over 3 hours once weekly. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients may also receive trastuzumab and/or pertuzumab per institution routine care per treating physician?s discretion.

ARM B: Patients receive docetaxel IV over 1 hour once every 3 weeks. Treatment repeats every 21 days for 4-6 cycles in the absence of disease progression or unacceptable toxicity. Patients may also receive cyclophosphamide, doxorubicin, trastuzumab, and/or pertuzumab per institution routine care per treating physician?s discretion.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be women with a known stage I-III invasive breast cancer diagnosis. Registration must occur within 84 days from the date of diagnosis
* Patients must be capable and willing to provide informed consent
* Patients must have plans to receive either neoadjuvant or adjuvant:

  * Every 3-week docetaxel x 4-6 cycles OR
  * Weekly paclitaxel x 4 cycles
  * NOTE: Recommended therapies for various therapy regimens are outlined based on estrogen receptor (ER)/progesterone receptor (PR)/HER2 and nodal status. Where there are options, the treating physician will choose a regimen best fitted for that patient. If the physician does not feel any of the regimens are the best fit for the patient, the patient should not be enrolled. Physicians will also document why a regimen was felt to be inappropriate when an option
* Patients must self-identify their race as black, African American, or of African descent; patients may be of any ethnicity
* Patients with a history of other cancers are eligible if they have not received prior taxane or platinum or vinca alkaloid therapy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Patients must not be pregnant or lactating

  * All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
  * A female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Women of childbearing potential must be strongly advised to use an accepted and effective method of contraception or to abstain from sexual intercourse for the duration of their participation in the study

Exclusion Criteria:

* Patients have received prior taxane or prior/concurrent platinum therapy
* Patients have pre-existing peripheral neuropathy
* Patients have a total bilirubin > upper limit of normal (ULN)
* Patients have aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) above 1.5 times the ULN concomitant with alkaline phosphatase above 2.5 times the ULN

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2027-03-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bryan P Schneider, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (485):
- United States (485):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Kingman Regional Medical Center, Kingman, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - PCR Oncology, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Cancer Center of Colorado at Sloan's Lake, Denver, Colorado
  - National Jewish Health-Main Campus, Denver, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - SCL Health Saint Joseph Hospital, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Good Samaritan Medical Center, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - McKee Medical Center, Loveland, Colorado
  - National Jewish Health-Northern Hematology Oncology, Thornton, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - SCL Health Lutheran Medical Center, Wheat Ridge, Colorado
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Suburban Hematology Oncology Associates - Snellville, Snellville, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Center, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of The Lake, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Our Lady of the Lake Physicians Group - Medical Oncology, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Woman's Hospital, Baton Rouge, Louisiana
  - Northshore Oncology Associates-Covington, Covington, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Saint Vincent Healthcare, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - The Cancer Institute of New Jersey Hamilton, Hamilton, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Inspira Medical Center Mullica Hill, Mullica Hill, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - South Carolina Cancer Specialists PC, Hilton Head Island, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Baptist Hospitals of Southeast Texas Cancer Center, Beaumont, Texas
  - Baptist Regional Cancer Network-Cancer Center of Southeast Texas, Port Arthur, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - Augusta Health Center for Cancer and Blood Disorders, Fishersville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Westchester Emergency Center, Midlothian, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Bon Secours Maryview Medical Center, Portsmouth, Virginia
  - Bon Secours Saint Mary's Hospital, Richmond, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Bon Secours Health Center at Harbour View, Suffolk, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Overlake Medical Center, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - MultiCare Gig Harbor Medical Park, Gig Harbor, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming

REFERENCES:
- [Derived] Schneider BP, Zhao F, Ballinger TJ, Garcia SF, Shen F, Virani S, Cella D, Bales C, Jiang G, Hayes L, Miller N, Srinivasiah J, Stringer-Reasor EM, Chitalia A, Davis AA, Makower DF, Incorvati J, Simon MA, Mitchell EP, DeMichele A, Miller KD, Sparano JA, Wagner LI, Wolff AC. ECOG-ACRIN EAZ171: Prospective Validation Trial of Germline Predictors of Taxane-Induced Peripheral Neuropathy in Black Women With Early-Stage Breast Cancer. J Clin Oncol. 2024 Aug 20;42(24):2899-2907. doi: 10.1200/JCO.24.00526. Epub 2024 Jun 3. PMID 38828938

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on June 27, 2019, first patient was enrolled on August 9, 2019. Accrual to arm A (paclitaxel) was terminated on June 4, 2021 and accrual to arm B (docetaxel) was terminated on March 31, 2022, after achieving the accrual goal on each arm separately.
Period: Overall Study
Arm/Group | Arm A (Paclitaxel) | Arm B (Docetaxel)
Started | 126 | 123
Received protocol therapy | 121 | 118
High Risk Genotype Group (Of the 121 treated patients on arm A, 4 patients did not have genotype data.) | 91 | 87
Low Risk Genotype Group | 26 | 31
Completed | 102 | 102
Not Completed | 24 | 21
Not completed — Never start protocol therapy | 5 | 5
Not completed — Adverse Event | 11 | 7
Not completed — Alternative therapy | 1 | 2
Not completed — Disease progression/relapse | 2 | 1
Not completed — Other complicating disease | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Ineligible | 2 | 2
Not completed — Reason missing due to delinquent data | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled to the trial
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Paclitaxel) | Arm B (Docetaxel) | Total
Number analyzed (Participants) | 126 | 123 | 249
Age, Continuous [Median (Full Range); unit: years] | 53 [23 to 72] | 56 [27 to 80] | 54 [23 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 123 | 249
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 121 | 118 | 239
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 125 | 123 | 248
  White | 0 | 0 | 0
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade 2-4 Taxane-Induced Peripheral Neuropathy (TIPN) by Genotype Risk Group in Arm A
Description: Grade 2-4 TIPN was assessed by treating physician using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. All patients who started protocol therapy on arm A (paclitaxel) were included in the analysis. The percentage of participants with grade 2-4 TIPN was calculated based on binomial distribution and was compared between high-risk vs low-risk genotype groups using Fisher exact test. Genotype risk group (high vs. low) was determined by genotyping. High-risk genotype was defined by FCAMR GG genotype (homozygous wild type) or SBF2 mutated. Low-risk genotype was defined by carriage of at least one variant allele in FCAMR (AG or AA) and SBF2 wild-type status.
Time Frame: assessed at baseline, an end of each cycle, at 6 months and 1 year post registration
Population: All patients on arm A who received at least one dose of paclitaxel and had genotyping results
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- High Risk Genotype Group: Germline neuropathy risk (high vs. low) was determined by genotyping. High-risk genotype was defined by FCAMR GG genotype (homozygous wild type) or SBF2 mutated.
- Low Risk Genotype Group: Germline neuropathy risk (high vs. low) was determined by genotyping. Low-risk genotype was defined by carriage of at least one variant allele in FCAMR (AG or AA) and SBF2 wild-type status.
Arm/Group | High Risk Genotype Group | Low Risk Genotype Group
Number analyzed (Participants) | 91 | 26
percentage of participants | 47 [38 to 56] | 35 [19 to 53]
Statistical Analysis 1: Comparison: High Risk Genotype Group vs Low Risk Genotype Group; Test type: Superiority; p = 0.27, Fisher Exact

2. Secondary Outcome: Patient-Reported Neuropathy Score Change Between Baseline and End of Treatment by Genotype Risk Group in Patients on Arm A
Description: The patient-reported neurotoxicity was assessed using the 11 items about neurotoxicity in the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity (FACT/GOG-Ntx) questionnaire (i.e., FACT/GOG-Ntx additional concerns subscale). The neurotoxicity total score was the sum of the scores for the 11 items, ranging from 0 to 44. Higher values of the FACT/GOG-Ntx neurotoxicity total score indicate less neurotoxicity. The FACT/GOG-Ntx neurotoxicity total score change between the baseline and at end of treatment (negative value indicates worsening symptom, positive value indicates improving symptom) was calculated and compared using two-sample t test. Genotype risk group (high vs. low) was determined by genotyping. High-risk genotype was defined by FCAMR GG genotype (homozygous wild type) or SBF2 mutated. Low-risk genotype was defined by carriage of at least one variant allele in FCAMR (AG or AA) and SBF2 wild-type status.
Time Frame: assessed at baseline and at end of treatment, an average of 3 months
Population: All patients who started paclitaxel and filled out the FACT/GOG-Ntx questionnaire at both baseline and end of treatment time points
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | High Risk Genotype Group | Low Risk Genotype Group
Number analyzed (Participants) | 81 | 24
score on a scale | -7.3 (9.1) | -8.1 (8.9)
Statistical Analysis 1: Comparison: High Risk Genotype Group vs Low Risk Genotype Group; Test type: Superiority; p = 0.96, t-test, 2 sided

3. Secondary Outcome: Percentage of Participants With Grade 2-4 TIPN Based on CTCAE Between Arm A and Arm B
Description: Grade 2-4 TIPN was assessed by treating physician using CTCAE version 4.0. All patients who started protocol therapy were included in the analysis. The percentage of participants with grade 2-4 TIPN was calculated based on binomial distribution and was compared between treatment arms using Fisher exact test.
Time Frame: assessed at baseline, an end of each cycle, at 6 months and 1 year post registration
Population: All patients who received at least one dose of protocol therapy
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Docetaxel)
Number analyzed (Participants) | 121 | 118
percentage of participants | 44 [36 to 52] | 25 [19 to 33]
Statistical Analysis 1: Comparison: Arm A (Paclitaxel) vs Arm B (Docetaxel); Test type: Superiority; p = 0.004, Fisher Exact

4. Secondary Outcome: Percentage of Participants With Dose Reduction Due to TIPN Between Arm A and Arm B
Description: The percentage of patients with dose reduction due to TIPN was calculated as number of patients with dose reduction due to peripheral neuropathy for any dose of any cycle divided by total number of patients who started protocol therapy. The percentages were calculated along with exact 95% CI based on binomial distribution and were compared between arms using Fisher exact test.
Time Frame: Dose reduction due to TIPN was assessed at end of each cycle, up to 4 cycles in arm A and 6 cycles in arm B
Population: All patients who received at least one dose of protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Docetaxel)
Number analyzed (Participants) | 121 | 118
percentage of participants | 28 [20 to 37] | 8 [4 to 15]
Statistical Analysis 1: Comparison: Arm A (Paclitaxel) vs Arm B (Docetaxel); Test type: Superiority; p < 0.001, Fisher Exact

5. Secondary Outcome: Percentage of Participants With Dose Reduction Due to Any Reason Between Arm A and Arm B
Description: The percentage of patients with dose reduction due to any reason was calculated as number of patients with any dose reduction for any dose of any cycle, regardless of the reason, divided by total number of patients who started protocol therapy. The percentages were calculated along with exact 95% CI based on binomial distribution and were compared between arms using Fisher exact test.
Time Frame: Dose reduction due to any reason was assessed at end of each cycle, up to 4 cycles in arm A and 6 cycles in arm B
Population: All patients who received at least one dose of protocol therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Paclitaxel) | Arm B (Docetaxel)
Number analyzed (Participants) | 121 | 118
percentage of participants | 39 [30 to 48] | 25 [17 to 33]
Statistical Analysis 1: Comparison: Arm A (Paclitaxel) vs Arm B (Docetaxel); Test type: Superiority; p = 0.019, Fisher Exact

6. Secondary Outcome: Percentage of Participants With Grade 2-4 TIPN by Genotype Risk Group in Arm B
Description: Grade 2-4 TIPN was assessed by treating physician using CTCAE version 4.0. All patients who started protocol therapy on arm B were included in the analysis. The percentage of participants with grade 2-4 TIPN was calculated based on binomial distribution and was compared between high-risk vs low-risk genotype groups using Fisher exact test. Genotype risk group (high vs. low) was determined by genotyping. High-risk genotype was defined by FCAMR GG genotype (homozygous wild type) or SBF2 mutated. Low-risk genotype was defined by carriage of at least one variant allele in FCAMR (AG or AA) and SBF2 wild-type status.
Time Frame: assessed at baseline, at end of each cycle, at 6 months and 1 year post registration
Population: All patients who received at least one dose of docetaxel and had genotyping results
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | High Risk Genotype Group | Low Risk Genotype Group
Number analyzed (Participants) | 87 | 31
percentage of participants | 28 [20 to 36] | 19 [9 to 35]
Statistical Analysis 1: Comparison: High Risk Genotype Group vs Low Risk Genotype Group; Test type: Superiority; p = 0.47, Fisher Exact

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle=21 days) while on treatment and for 30 days after the end of treatment, then at 6 months, 1, 2 and 3 years post registration
Description: All patients are included in the all-cause mortality analysis and only treated patients are included in the AE analysis
Arm/Group | Arm A (Paclitaxel) | Arm B (Docetaxel)
All-Cause Mortality (participants affected / at risk) | 7/126 | 6/123
Serious Adverse Events (participants affected / at risk) | 46/121 | 61/118
Other Adverse Events (participants affected / at risk) | 121/121 | 113/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Paclitaxel) (N=121) | Arm B (Docetaxel) (N=118)
Anemia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1
Blood and lymphatic system disorders -Other (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Chest pain - cardiac (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1
Right ventricular dysfunction (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Cardiac disorders - Other (Cardiac disorders) | 1 | 1
Chills (General disorders and administration site conditions) | 0 | 1
Edema limbs (General disorders and administration site conditions) | 3 | 3
Fatigue (General disorders and administration site conditions) | 1 | 2
Fever (General disorders and administration site conditions) | 1 | 3
Flu like symptoms (General disorders and administration site conditions) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Non-cardiac chest pain (General disorders and administration site conditions) | 0 | 3
Pain (General disorders and administration site conditions) | 2 | 1
Disease progression (General disorders and administration site conditions) | 0 | 1
Generalized edema (General disorders and administration site conditions) | 0 | 1
General disorders and administration site conditions - Other (General disorders and administration site conditions) | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Anal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 5 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 9
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 5
Nausea (Gastrointestinal disorders) | 2 | 10
Stomach pain (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 6
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 4
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 2
Anaphylaxis (Immune system disorders) | 0 | 1
Immune system disorders - Other (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Breast infection (Infections and infestations) | 0 | 1
Laryngitis (Infections and infestations) | 0 | 2
Lung infection (Infections and infestations) | 1 | 1
Rash pustular (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 3
Tracheal obstruction (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Creatinine increased (Investigations) | 1 | 2
Neutrophil count decreased (Investigations) | 1 | 4
Platelet count decreased (Investigations) | 1 | 3
Urine output decreased (Investigations) | 0 | 1
Weight loss (Investigations) | 1 | 1
White blood cell decreased (Investigations) | 0 | 3
Investigations - Other (Investigations) | 2 | 2
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Neuralgia (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 4 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 15
Stroke (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Watering eyes (Eye disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 0 | 1
Hematoma (Vascular disorders) | 1 | 0
Hot flashes (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Paclitaxel) (N=121) | Arm B (Docetaxel) (N=118)
Anemia (Blood and lymphatic system disorders) | 70 | 71
Edema limbs (General disorders and administration site conditions) | 8 | 18
Fatigue (General disorders and administration site conditions) | 64 | 75
Pain (General disorders and administration site conditions) | 24 | 18
General disorders and administration site conditions - Other (General disorders and administration site conditions) | 6 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 32 | 51
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 9
Nail discoloration (Skin and subcutaneous tissue disorders) | 15 | 21
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 14
Rash acneiform (Skin and subcutaneous tissue disorders) | 6 | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 13 | 16
Nail changes (Skin and subcutaneous tissue disorders) | 16 | 13
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 7
Abdominal pain (Gastrointestinal disorders) | 11 | 5
Constipation (Gastrointestinal disorders) | 23 | 30
Diarrhea (Gastrointestinal disorders) | 29 | 48
Dyspepsia (Gastrointestinal disorders) | 6 | 11
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 6
Mucositis oral (Gastrointestinal disorders) | 13 | 18
Nausea (Gastrointestinal disorders) | 34 | 45
Vomiting (Gastrointestinal disorders) | 11 | 11
Infections and infestations - Other (Infections and infestations) | 3 | 6
Alanine aminotransferase increased (Investigations) | 21 | 11
Alkaline phosphatase increased (Investigations) | 8 | 5
Aspartate aminotransferase increased (Investigations) | 12 | 8
Creatinine increased (Investigations) | 6 | 13
Lymphocyte count decreased (Investigations) | 33 | 13
Neutrophil count decreased (Investigations) | 22 | 14
Platelet count decreased (Investigations) | 5 | 7
White blood cell decreased (Investigations) | 46 | 30
Investigations - Other (Investigations) | 6 | 12
Anorexia (Metabolism and nutrition disorders) | 13 | 26
Hyperglycemia (Metabolism and nutrition disorders) | 33 | 35
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 | 13
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 11
Hypokalemia (Metabolism and nutrition disorders) | 14 | 18
Hyponatremia (Metabolism and nutrition disorders) | 7 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 20
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 14
Dizziness (Nervous system disorders) | 10 | 15
Dysgeusia (Nervous system disorders) | 7 | 19
Headache (Nervous system disorders) | 20 | 27
Paresthesia (Nervous system disorders) | 7 | 5
Peripheral motor neuropathy (Nervous system disorders) | 26 | 26
Peripheral sensory neuropathy (Nervous system disorders) | 112 | 91
Blurred vision (Eye disorders) | 5 | 11
Anxiety (Psychiatric disorders) | 15 | 14
Depression (Psychiatric disorders) | 6 | 10
Insomnia (Psychiatric disorders) | 20 | 21
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 21 | 23
Breast pain (Reproductive system and breast disorders) | 7 | 10
Hot flashes (Vascular disorders) | 17 | 24
Hypertension (Vascular disorders) | 21 | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/29/NCT04001829/Prot_SAP_000.pdf